CLINICAL TRIAL: NCT01329835
Title: Effect of Psycho-education on Gestational Weight Gain and Anxiety/Depression in Obese Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Limburg Catholic University College (Other)
Collaborators: PHL University College (Unknown)
Responsible Party: Wim Jackmaer, PHL University College
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GWG32011
Record Dates: First submitted 2011-03-30; First posted 2011-04-06 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2008-07

CONDITIONS: Obese Pregnant Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Written information via brochure (Experimental): Written information by a brochure
  Interventions: Other: brochure
- standard care (No Intervention): standard prenatal care
- Lifestyle counseling (Experimental): Psycho-education based on principles of motivational interviewing and positive reinforcement
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: Lifestyle counseling — 4 prenatal sessions based on principles of motivational interviewing and positive reinforcement
  Arms: Lifestyle counseling
Other: brochure — brochure given after randomization
  Arms: Written information via brochure

SUMMARY:
Prepregnancy obesity, defined as a body mass index (BMI) of 30kg/m² or more, shows a strong association with pregnancy and birth complications for both the mother and her child. Most consequently reported maternal risks include an increased risk for gestational diabetes, hypertension and pre-eclampsia, increased incidence of induction of labour, operative delivery, postpartum haemorrhage, anaesthetic risks as well as risk for infections and thromboembolic complications. Fetal risks include miscarriage, neural-tube defects, heart defects, macrosomia and stillbirth. Initiation and continuation of breastfeeding is more complicated in obese women than in normal weight women. Also in later life chronic diseases can put the mother and her baby's health at risk. The Institute Of Medicine (IOM) guidelines suggest a gestational weight gain (GWG) to be limited to 5 - 9 kg (11-19,8 lb) in obese women in order to minimize the synergetic negative health consequences of excessive weight gain for both the obese mother and her child. Preventing excessive weight gain during pregnancy and postpartum weight retention is also important in the prevention of overweight and obesity among women of reproductive age. Obese women in general have a poor diet quality and are more exposed to psychosocial factors like anxiety and feelings of depression than normal weight women.

The aim of this project is to perform a randomized controlled trial (RCT) in order to evaluate the effects of life-style intervention (psycho-education by a midwife during 4 prenatal sessions) on pregnancy and birth outcomes. Main dependent variables are gestational weight gain and anxiety and depression. Obesity is a modifiable risk factor and optimizing an adequate gestational weight gain with attention to psycho-social factors, can reduce the need for adverse perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Less than 15 weeks pregnant

Exclusion Criteria:

* Multiple pregnancy
* Preexisting diabetes
* Primary need for nutritional advice
* Inadequate knowledge of Dutch language

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2008-03; Primary Completion 2011-04 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Gestational weight gain | For the duration of pregnancy, an expected average of 40 weeks
  Weight just before delivery minus prepregnancy weight

SECONDARY OUTCOMES:
Evolutions in anxiety and depression during pregnancy | During pregnancy on fixed time points: trimester 1 (before 15 weeks of gestation), trimester 2 (between 18 and 28 weeks of gestation) and trimester 3 (between 30 - 34 weeks of gestation)
  STAI (Spielberger) ==> anxiety EPDS ==> depression

CONTACTS AND LOCATIONS:
Overall Officials: Roland Devlieger, PhD, MD, Study Director — Universitaire Ziekenhuizen KU Leuven; Bea Van den Bergh, PhD, Study Director — University of Tilburg (Nl); Ingrid Witters, PhD, MD, Study Director — Universitaire Ziekenhuizen KU Leuven; Annick Bogaerts, MW, MSc, PhDstudent, Principal Investigator — KHLim PHL
Locations (3):
- Belgium (3):
  - St-Jans Hospital ZOL, Genk, Limburg
  - Jessa Hospital, Hasselt, Limburg
  - SFZ, Heusden, Limburg